CLINICAL TRIAL: NCT01636453
Title: The Penumbra Liberty Trial: Safety and Effectiveness in the Treatment of Wide-Neck Intracranial Aneurysms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP 5038 (IDE # G120050)
Record Dates: First submitted 2012-07-02; First posted 2012-07-10 (Estimated); Results first posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-04

CONDITIONS: Wide-neck, Saccular Intracranial Aneurysms
Keywords: wide-neck; saccular; intracranial aneurysms; ICA; Stent assisted coiling; Liberty Stent
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liberty Stent arm (Experimental): Patients are implanted with the Liberty Stent as an assist to embolic coiling of their wide-neck, saccular, intracranial aneurysms and follow for 12 months
  Interventions: Device: Stent assisted coiling with the Liberty Stent

INTERVENTIONS:
Device: Stent assisted coiling with the Liberty Stent — Patients are implanted with the Liberty Stent as an assist to embolic coiling of their wide-neck, saccular, intracranial aneurysms and follow for 12 months

SUMMARY:
To assess the safety and effectiveness of the Penumbra Liberty Stent System as adjunctive treatment to embolic coils for wide-neck, saccular, intracranial aneurysms in the internal carotid artery (ICA). The Liberty Stent System is an implantable device comprised of a stent and delivery system designed as an adjunct to embolic coils in the treatment of wide-neck, saccular, intracranial aneurysms. It has three components: an implant, an introducer sheath and a delivery wire assembly. The implant component is made of superelastic and biocompatible nitinol tubular material. Patients presenting with wide-neck, saccular, intracranial aneurysms in the internal carotid artery (ICA) from the cavernous segment to the carotid terminus (including the paraclinoid, ophthalmic, hypophyseal and posterior communicating segments) will receive stent assisted coiling by the Penumbra Liberty Stent with any approved embolic coils currently on the market. Wide-neck aneurysms are defined by a neck ≥4mm or a dome-to-neck ratio <2. Each patient will be followed and assessed for 2, 6 and 12 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* A wide-neck intracranial saccular aneurysm with a neck ≥ 4mm or a dome to neck ratio <2 in the ICA from the cavernous segment to the carotid terminus (including the paraclinoid, ophthalmic, hypophyseal and posterior communicating segments)
* Life expectancy > 12 months
* Signed Informed Consent

Exclusion Criteria:

* Females who are pregnant or intend to become pregnant during the study. (Females of child-bearing potential must have a urinary pregnancy test within 7 days of enrollment)
* Extradural aneurysms
* Known multiple untreated cerebral aneurysms at study entry
* Recent history of subarachnoid hemorrhage, intracranial hemorrhage, or major surgery within one month of enrollment
* Admission platelet <50,000 or any known hemorrhagic diathesis, coagulation deficiency, or on oral anticoagulant therapy with an INR >3.0
* Contraindication to angiography such as elevated creatinine or known allergy to angiographic contrast
* Contraindication to CT and/or MRI scans
* Known allergy to the metal component of the Penumbra Liberty Stent System
* Evidence of active infection (WBC >10x109 /L)
* Any medical conditions that will not allow the necessary follow-up for this study (e.g., pre-existing neurological or psychiatric diseases)
* Current substance-abuse /illicit drug use
* Angiographic evidence of an arterial stenosis proximal to the target lesion that could prevent device deployment
* Contraindications to study medications (heparin, aspirin, clopidogrel, and radiographic contrasts)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Demtrius Lopes, MD, Principal Investigator — Rush University Medical Center; Henry Woo, MD, Principal Investigator — Stony Brook University Medical Center
Locations (3):
- United States (3):
  - Swedish Medical Center, Denver, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Stony Brook University Medical Center, Stony Brook, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liberty Stent Arm
Started | 120
Completed | 112
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Liberty Stent Arm
Number analyzed (Participants) | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 78
  >=65 years | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 27
  Race: Black | 17
  Race: Caucasian | 61
  Race: American Indian | 1
  Race: Other | 2
  Race: Unknown | 4
Region of Enrollment [Number; unit: participants]
  United States | 95
  Japan | 25
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 26.9 [23.4 to 32]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Raymond Class I Complete Obliteration at 12 Months
Description: Complete aneurysmal obliteration is defined by the method of Raymond et al. (Class I) (Stroke 2001;32:1998-2004).
Time Frame: At 12 months post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Liberty Stent Arm
Number analyzed (Participants) | 109
Participants | 98

2. Primary Outcome: Number of Neurological Deaths or Major Ipsilateral Strokes at 12 Months Post Treatment.
Time Frame: At 12 months post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Liberty Stent Arm
Number analyzed (Participants) | 112
Participants | 3

3. Secondary Outcome: Number of Ipsilateral Ischemic Strokes
Description: Defined as episodes of focal or global neurological dysfunction due to brain or retinal infarction in the same hemisphere of the target aneurysm with signs and symptoms that persist for 24 hours or longer. When appropriate, non contrast CT scans will be used to eliminate hemorrhagic strokes
Time Frame: At 12 months post-implant
Measure: Number; unit: participants
Arm/Group | Liberty Stent Arm
Number analyzed (Participants) | 112
participants | 8

4. Secondary Outcome: Number of Participants With Device-related Serious Adverse Events
Description: The number of participants with device-related Serious Adverse Events as a measure of safety of the procedure and device. The FDA definitions for Serious Adverse Events are used.
Time Frame: During the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Liberty Stent Arm
Number analyzed (Participants) | 112
Participants | 17

5. Secondary Outcome: Number of Device Deployment Failures
Description: Defined by the failure of the device to deploy or failure to correctly position the device over the aneurysm
Time Frame: During the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Liberty Stent Arm
Number analyzed (Participants) | 112
Participants | 5

6. Secondary Outcome: Number of Device Migrations
Description: Migration is defined as movement of the Liberty stent by more than 5 mm as documented by the 12 month angiogram when compared to its immediate post-implant position.
Time Frame: 12 months post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Liberty Stent Arm
Number analyzed (Participants) | 105
Participants | 0

7. Secondary Outcome: Number of Participants With Aneurysm Raymond Class I Occlusion Grading
Description: Raymond Class I Occlusion grading defined as complete obliteration of the aneurysm at 12 months.
Time Frame: At 12 months post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Liberty Stent Arm
Number analyzed (Participants) | 109
Participants | 99

8. Secondary Outcome: Number of Intracranial Hemorrhages
Description: Inclusive of subarachnoid, intraventricular or intraparenchymal hemorrhages (symptomatic or asymptomatic). Symptomatic is defined as a 4 point or more increase in the National Institutes of Health Stroke Scale (NIHSS) from baseline. The NIHSS ranges from 1 to 42, with higher scores indicating greater severity of stroke.
Time Frame: At 12 months post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Liberty Stent Arm
Number analyzed (Participants) | 112
Participants | 2

9. Secondary Outcome: Number of Participants With Functional Outcome as Defined by the Modified Rankin Scale (mRS) 0-2
Description: The Modified Rankin Scale measures functional ability on a scale from 0-5, with 0 indicating no symptoms at all and 5 indicating severe disability.
Time Frame: At 12 months post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Liberty Stent Arm
Number analyzed (Participants) | 107
Participants | 106

10. Secondary Outcome: All Cause Mortality (Number of Deaths From Any Cause)
Time Frame: At 12 months post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Liberty Stent Arm
Number analyzed (Participants) | 112
Participants | 0

11. Secondary Outcome: Number of Retreatments
Description: Defined as any intervention after the completion of the initial stent assisted coiling procedure
Time Frame: At 12 months post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Liberty Stent Arm
Number analyzed (Participants) | 112
Participants | 4

12. Secondary Outcome: Number of Participants Who Experienced Device Patency
Description: Device patency (stenosis) at 12 months
Time Frame: at 12 months post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Liberty Stent Arm
Number analyzed (Participants) | 105
Participants | 2

13. Secondary Outcome: Number of Participants Who Experienced Aneurysm Recanalization
Time Frame: At 12 months post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Liberty Stent Arm
Number analyzed (Participants) | 112
Participants | 6

ADVERSE EVENTS:
Arm/Group | Liberty Stent Arm
Serious Adverse Events (participants affected / at risk) | 34/112
Other Adverse Events (participants affected / at risk) | 96/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liberty Stent Arm (N=112)
Nervous System Disorders (Nervous system disorders) | 19
Infections and Infestations (Infections and infestations) | 7
Gastrointestinal Disorders (Gastrointestinal disorders) | 6
General Disorders (General disorders) | 6
Cardiac Disorders (Cardiac disorders) | 3
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 3
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 2
Eye Disorders (Eye disorders) | 2
Neoplasms, benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Vascular Disorders (Vascular disorders) | 2
Hepatobiliary Disorders (Hepatobiliary disorders) | 1
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1
Psychiatric Disorders (Psychiatric disorders) | 1
Respiratory, Thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liberty Stent Arm (N=112)
Nervous System Disorders (Nervous system disorders) | 60
General Disorders (General disorders) | 23
Infections and Infestations (Infections and infestations) | 22
Eye Disorders (Eye disorders) | 34
Vascular Disorders (Vascular disorders) | 15
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 12
Injury, poisoning, and procedural complications (Injury, poisoning and procedural complications) | 11
Muskuloskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 10
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 9
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 6
Cardiac disorders (Cardiac disorders) | 6
Immune System Disorders (Immune system disorders) | 6
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 6
Renal and urinary disorders (Renal and urinary disorders) | 6
Ear and labyrinth disorders (Ear and labyrinth disorders) | 4
Investigations (Investigations) | 2
Reproductive system and breast disorders (Reproductive system and breast disorders) | 2
Endrocrine disorders (Endocrine disorders) | 1
Psychiatric Disorders (Psychiatric disorders) | 1
Surgical and Medical Procedures (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No